CLINICAL TRIAL: NCT03383835
Title: Feasibility Study of Moderate Dose Omega 3 Fatty Acid Supplementation in Premenopausal Women at High Risk for Breast Cancer Considering Future Pregnancy
Brief Title: Study of Moderate Dose Omega 3 Fatty Acid Supplement in Premenopausal Women at High Risk for Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lauren Nye (Other)
Collaborators: University of Kansas Medical Center (Other); American Cancer Society, Inc. (Other)
Responsible Party: Sponsor-Investigator, Lauren Nye, Medical Doctor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Moderate Dose Omega-3
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
Keywords: Omega 3 supplement; pre-menopausal; pregnancy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Omega-3 Supplementation (Experimental): Participants will take the dose of omega-3 supplementation (600mg DHA and 300mg EPA) daily for 6 months.
  Interventions: Dietary Supplement: Omega-3 Supplementation

INTERVENTIONS:
Dietary Supplement: Omega-3 Supplementation — DHA 600 milligrams (mg) per day for 6 months
  EPA 300mg per day for 6 months

SUMMARY:
This pilot study is an investigation of feasibility of moderate dose omega-3 fatty acid supplementation in pre-menopausal women at high risk for breast cancer who are considering future pregnancy. The goal of this pilot study is to determine feasibility of the study, document compliance with omega-3 fatty acid supplementation in this population and identify novel biomarkers modulated by moderate dose omega-3 fatty acids in this population.

DETAILED DESCRIPTION:
Pregnancy and breast feeding are protective when they occur at an early age, typically at an age less than 30. The influence of pregnancy on breast cancer risk is not fully understood, and little is known about modulation of the breast microenvironment during pregnancy and its influence on risk. Hormones, including rising estrogen levels, play a role in fatty acid synthesis. In pre-clinical models, a rise in omega-3:omega-6 ratio occurs naturally in the breast of pregnant mice. This may be able to be accentuated in human breast tissue with omega-3 fatty acid supplementation. Omega-3 fatty acid supplementation has been shown to favorably modulate breast cancer risk and risk biomarkers in pre-menopausal women at high risk for breast. Omega-3 fatty acid supplementation during pregnancy has also been found to have positive outcomes for the offspring, making it an ideal intervention to study in this population.

This pilot study of omega-3 supplementation in pre-menopausal women at high risk for breast cancer who are still considering pregnancy is addressing a potential prevention strategy in a population otherwise excluded from breast cancer prevention trials and not eligible for standard of care chemoprevention. With this pilot, the intent is to establish feasibility, document tolerability, determine number of women needed to enroll based on pregnancy rate and identify biomarkers for future investigation. This information will provide necessary data to apply for future extramural funding for a larger randomized trial. In a larger randomized trial with longer follow up, we will be able to assess post-pregnancy breast tissue and biomarkers to examine efficacy of omega-3 fatty acid supplementation in breast cancer risk reduction.

ELIGIBILITY:
Inclusion Criteria:

* Women age 21 - 40 must be pre-menopausal as defined as having intact ovaries with regular menses or if not menstruating, have a premenopausal status confirmed by serum follicle-stimulating hormone (FSH) and estradiol.
* Women must be considered at high risk for breast cancer based on family history (first or second degree relative diagnosed with breast cancer under the age of 60), prior precancerous biopsy or a 5-year Gail model risk estimate of ≥ 1.7% or 10 year Tyrer-Cuzick risk of 2x population risk as listed in the model.
* Women must indicate that they are still considering future pregnancy and childbearing.
* Women must be one year from pregnancy and breast-feeding.
* Women must be willing to take supplemental omega-3 fatty acids provided by the study.

Exclusion Criteria:

* Women actively undergoing in-vitro fertilization or fertility treatments are excluded.
* Women currently pregnant or breast-feeding at time of study consent.
* Women with an active malignancy.
* Women on anticoagulation.
* Women with bilateral breast implants or tram flap reconstruction.
* Women who have had radiation to both breasts.
* Women with current mammographic or clinical breast exam mass which is suspicious for breast cancer and malignancy has not been ruled out.

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Follow-up visit completion rate | 6 months
  Defined as the overall completion of 80% of follow-up visits study-wide.

SECONDARY OUTCOMES:
Pregnancy rate | 6 months
  Pregnancy will be assessed by review of patient record.
Discontinuation rate of omega-3 supplementation | 6 months
  Discontinuation rate will be assessed by patient reported compliance.
Incidence of microbiome in collected breast tissue | 6 months
  Microbiome will be assessed with random periareolar fine-needle aspiration (RPFNA)
Identify presence of biomarkers | 6 months
  Biomarkers will be assessed by RPFNA

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Nye, MD, Principal Investigator — The University of Kansas - Cancer Center
Locations (1):
- The University of Kansas Cancer Center, Westwood, Kansas, United States